CLINICAL TRIAL: NCT02460393
Title: A Randomized, Double Blind, Placebo Controlled Trial With Humanized TNFα Monoclonal Antibody Injection by Single Dose and Dose Escalation to Explore the Tolerance, Safety and Pharmacokinetic Characteristics in Healthy Subjects
Brief Title: A Trial With Humanized TNFα Monoclonal Antibody Injection by Single Dose and Dose Escalation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sss07
Record Dates: First submitted 2015-01-18; First posted 2015-06-02 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Rheumatoid Arthritis
Keywords: tolerance; safety and pharmacokinetic characteristics
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): The arm is as a control group to study the tolerance, safety and pharmacokinetic characteristics of Subcutaneous injection of different doses of humanized TNFα monoclonal antibody.
  Interventions: Other: placebo
- experimental group (Experimental): The arm is as an experimental group to study the tolerance, safety and pharmacokinetic characteristics of Subcutaneous injection of different doses of humanized TNFα monoclonal antibody.
  Interventions: Drug: Humanized TNFα monoclonal antibody

INTERVENTIONS:
Drug: Humanized TNFα monoclonal antibody — Subcutaneous injection of different doses for healthy people
  Subcutaneous injection of different doses in healthy people
  Other Names: TNFα monoclonal antibody
  Arms: experimental group
Other: placebo — Subcutaneous injection of different doses for healthy people
  Arms: Placebo group

SUMMARY:
This study is a randomized, double-blind and placebo-controlled trial with healthy subjects. There are 6 Groups as follows: 5mg, 15mg, 30mg, 50mg, 75mg, 100mg, and each group includes12 people. A single subcutaneous injection will be administrated starting from the low dose group (in accordance with 5mg, 15mg, 30mg, 50mg, 75mg, 100mg administered subcutaneously). Pharmacokinetics and pharmacodynamics data will be collected; drug metabolism and pharmacokinetics characteristics will be analyzed. Drug safety and tolerance for subjects will be evaluated.

DETAILED DESCRIPTION:
This study is a randomized, double-blind and placebo-controlled trial with healthy subjects. There are 6 Groups as follows: 5mg, 15mg, 30mg, 50mg, 75mg, 100mg, and each group includes12 people. A single subcutaneous injection will be administrated starting from the low dose group (in accordance with 5mg, 15mg, 30mg, 50mg, 75mg, 100mg administered subcutaneously). Pharmacokinetics and pharmacodynamics data will be collected; drug metabolism and pharmacokinetics characteristics will be analyzed. Drug safety and tolerance for subjects will be evaluated.

The study observed blood concentrations of the experimental drug at different time points after and before administration, TNFα before and after treatment at different time points will be observed as well.

C-T curve will be drawn with blood drug concentration (c) and time (T) in the trial. At the same time, the investigators will draw the average plasma concentration curve. Compartmental and non compartmental model will be used to analyze the pharmacokinetic parameters of subjects. It will be judged with linear or nonlinear elimination by the correlation analysis of AUC, Cmax of different doses. In the meantime, adverse events, vital signs, physical examination, laboratory examination and ECG will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adult volunteers who are voluntary to participate in clinical trials, and signed the informed consent
2. aged 18-45 years, the same batch of subjects age difference is less than or equal to 10 years of age
3. subjects with qualified physical examination within 7 days before the trial, body mass index (BMI) from19 to 24 ,and the same batch of subjects are with the similar weight
4. the basic indicators of heart, liver, kidney and blood examination are in the normal range.

Exclusion Criteria:

1. subjects are during the acute or chronic infection period, or have a previous history of active tuberculosis
2. subjects are with the history of diseases of the central nervous system, cardiovascular system, kidney, liver (specific indexes of liver function), digestive system ,respiratory system or metabolic system or suffered from other significant disease
3. subjects as allergic constitution after inquiry, suspected or confirmed or have a history of drug, food allergy , or subjects with a clear history of allergies and / or allergic to the humanized TNF alpha monoclonal antibody or the ingredient of humanized TNF alpha monoclonal antibody , or serum immunoglobulin E (IgE) examination was abnormal
4. subjects are included in other clinical trials of other drugs 3 months before being enrolled in this clinical trial, or candidates used drugs known to have damage to the main organs within 3 months before this trial;
5. candidates with blood donation history 3 months before being enrolled
6. Prescription and non prescription drugs were administrated Within 2 weeks before inclusion
7. ALT or AST > 1.5N (the upper limit of normal), Cr>N (the upper limit of normal);
8. leukocyte absolute value less than 3.50 × 109/L or > 9.50× 109/L, neutrophil absolute value less than 1.8× 109/L, platelet counts less than 100 × 109/L, hemoglobin is less than 100g/L
9. hepatitis B surface antigen (HbsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome (Anti-HIV) antibody and anti Treponema pallidum antibody (TP-Ab) are positive subjects
10. candidates with positive tuberculin skin test with 5 unit dose tuberculin , the size of 48-72 hour scleroma greater than 5 mm
11. subjects with positive anti nuclear antibodies (ANA, ds-DNA, ENA)
12. subjects with positive resistantance antibody
13. subjects had a history of mental illness
14. subjects who are pregnant, lactating women or a planning pregnant within 3 months
15. subjects with the history of orthostatic hypotension
16. with drug or drug abuse history after inquiry
17. daily smoking more than 5 cigarettes or the same amount of tobacco after inquiry
18. subjects drink more than 28 units of alcohol after inquiry, or alcohol breath test are positive within 24 hours before the acceptance of the tested drugs
19. There is a family history of cancer
20. Significantly abnormal values in clinical appeared during the screening
21. subjects cannot understand, exchangeand cooperate enough, and cannot guarantee the researchers according to the scheme
22. researchers don't think it is right to participate in the research with other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
AUC | 28 days
  AUC
Cmax | 28 days
  Cmax
Cmin | 28 days
  Cmin
Tmax | 28 days
  Tmax

SECONDARY OUTCOMES:
Serum creatinine and AST and ALT | 28 days
  Serum creatinine and AST and ALT
or any other adverse events | 28 days
  or any other adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China